CLINICAL TRIAL: NCT06447649
Title: Investigation of Factors Affecting Shoulder Pain in Stroke Survivors
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Emre BASKAN, Associate Professor, Pamukkale University
Other Study IDs: PAU-FTR-CA-01
Record Dates: First submitted 2024-05-31; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Stroke
Keywords: Functionality; Hemiplegic Shoulder Pain; Stroke; Muscle Tone; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: We included stroke patients aged between 20 and 85. inclusion criteria for this study; having received a diagnosis of hemiplegia following a cerebrovascular accident (CVA), having experienced a first-time stroke, having unilaterally affected, having stage 3 or above Brunnstrom upper limb stage, not having any other neurological/orthopedic problems in addition to hemiplegia, not having any shoulder problems on the same side (affected side) before the stroke, scoring 25 or above on the Mini Mental Test.

SUMMARY:
The aim of this study was to examine the factors affecting shoulder pain in stroke survivors and to determine how much the factors affect shoulder pain

DETAILED DESCRIPTION:
The study included 62 stroke patients who got stage 3 or more from the Brunnstrom upper limp stage. We assessed shoulder pain using the Visual Analog Scale, evaluated muscle tone using the Modified Ashworth Scale, identified myofascial trigger points by manual palpation, and measured range of motion using a universal goniometer. We employed the Fugl-Meyer Upper Extremity Assessment to assess the functional status of the upper extremities. We also used the Neer Impingement, Apprehension, Acromioclavicular Shear, and Speed Tests to evaluate the soft tissue condition.

ELIGIBILITY:
inclusion Criteria:

* having received a diagnosis of hemiplegia following a cerebrovascular accident (CVA)
* having experienced a first-time stroke
* having unilaterally affected, having stage 3 or above Brunnstrom upper limb stage
* not having any other neurological/orthopedic problems in addition to hemiplegia
* not having any shoulder problems on the same side (affected side) before the stroke
* not having any shoulder problems on the same side (affected side) before the stroke

Exclusion Criteria:

* having a history of shoulder injury (affected side)
* neurological and orthopedic diseases other than stroke
* prior stroke
* bilateral involvement
* non-cooperation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stroke patients treated in the Physical Therapy and Rehabilitation Unit of Pamukkale University Faculty of Medicine Hospital. We conducted patient selection through screening using the Probel system, and randomly assigned patients who met the inclusion criteria and agreed to participate in the study using a random number table.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 1 year
  Visual Analog Scale (VAS) used to asses shoulder pain of stroke survivors. The patient will be asked to indicate the point on a 10 cm line that best represents their pain, with 0 indicating no pain and 10 indicating unbearable pain. Subsequently, the distance of the point from the 0 point will be measured using a ruler to determine the intensity of the pain. Following this, the patient will be inquired about the localization and type of pain.
Modified Ashworth Scale (MAS) | 1 year
  Modified Ashworth Scale (MAS) used to evaluated of muscle tone. A scale commonly used for spasticity assessment in clinical settings. The initial form, known as the Ashworth Scale, categorizes the resistance of the extremity to passive movement within a range of 0-4 points. Subsequently, the scale includes a value of 1+, defining it as the 6-point Modified Ashworth Scale. (9) According to MAS
Fugl Meyer Motor Assesment Scale (FMMAS) | 1 year
  Fugl Meyer Motor Assesment Scale (FMMAS) was employed to evaluate motor recovery after a stroke, it is a disease-specific, reliable, and up-to-date scale. It includes sub-sections assessing joint movements, coordination, and reflex activities related to the shoulder, elbow, forearm, wrist, and hand. The maximum score achievable from the upper extremity assessment is 66,
Neer Impingement Test | 1 year
  Neer Impingement Test was used to identify possible subacromial impingement syndrome. The patient's shoulder is passively brought into flexion and internal rotation position. The positive examination finding is the occurrence of shoulder pain during the movement of the arm in this position. The test has a sensitivity of 68% and a specificity of 68.7%.
Speed Test | 1 year
  Speed Test was used to identify possible biceps tendon pathologies. When shoulder flexion is performed against resistance with the elbow extended and the forearm supinated, the presence of pain in the bicipital groove indicates a positive test.
Acromioclavicular Shear Test | 1 year
  Acromioclavicular Shear Test was used to identify acromioclavicular joint pathology. The examiner cups their hands over the shoulder with the heel of one hand on the clavicle, and the heel of the other on the spine of the scapula, and then squeeze their hands together. A positive result is abnormal movement or pain at the acromioclavicular joint. The test has a sensitivity of 100% and a specificity of 97%
Apprehension Test | 1 year
  Apprehension Test was used to detect the presence of anterior instability. As the shoulder is passively moved into maximum external rotation in abduction, and forward pressure is applied to the posterior aspect of the humeral head. If the patient expresses concern about dislocation or reports pain in the shoulder, the test is considered positive. The test has a sensitivity of 58% and a specificity of 96%

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No